CLINICAL TRIAL: NCT01462318
Title: A Multicenter, Single-Arm, Open-Label Study to Evaluate the Immunogenicity and Pharmacokinetics of BIIB019, Daclizumab High Yield Process (DAC HYP), Prefilled Syringe Administered by Subcutaneous Injection in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: An Open-Label Immunogenicity and Pharmacokinetics Study of Daclizumab High Yield Process Prefilled Syringe in Relapsing Remitting Multiple Sclerosis
Acronym: OBSERVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 205MS302; 2010-023856-97 (EudraCT Number)
Record Dates: First submitted 2011-07-14; First posted 2011-10-31 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Pre-filled syringe; Pharmacokinetic; Daclizumab High Yield Process; immunogenicity
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Midazolam; Caffeine; Warfarin; Vitamin K; Omeprazole; Dextromethorphan; Daclizumab; daclizumab HYP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DAC HYP (Experimental): DAC HYP 150 mg by a subcutaneous (SC) injection using the pre-filled syringe (PFS) every 4 weeks for 24 weeks followed by a 20-week washout period. After completion of the washout period, participants may resume monthly DAC HYP 150 mg using the PFS for up to 3 additional years.
  Participants in the TP-DI sub-study will receive probe-drug cocktail administration at Weeks 43 and 53. The probe-drug cocktail consists of oral midazolam 5 mg, caffeine 200 mg, S-warfarin 10 mg, vitamin K 10 mg, omeprazole 40 mg, and dextromethorphan 30 mg. The oral vitamin K is used to counteract warfarin's anticoagula nt effect prophylactically.
  Interventions: Drug: Midazolam; Other: Caffeine; Drug: S-warfarin; Other: Vitamin K; Drug: Omeprazole; Drug: Dextromethorphan; Biological: BIIB019 (Daclizumab)

INTERVENTIONS:
Drug: Midazolam — 5 mg
Other: Caffeine — 200 mg
Drug: S-warfarin — 10 mg
Other: Vitamin K — 10 mg
Drug: Omeprazole — 40 mg
Drug: Dextromethorphan — 30 mg
Biological: BIIB019 (Daclizumab) — 150 mg in 1 ml PFS
  Other Names: Daclizumab High Yield Process; DAC HYP

SUMMARY:
The primary objective of the study is to assess the immunogenicity of Daclizumab High Yield Process (DAC HYP) 150 mg administered every 4 weeks by subcutaneous (SC) injection using the pre-filled syringe (PFS) in participants with relapsing-remitting multiple sclerosis (RRMS). The secondary objectives of this study are to characterize the pharmacokinetics (PK) of DAC HYP following single and multiple doses of DAC HYP administered by the PFS in a subset of participants with RRMS and to evaluate the effect of DAC HYP on the PK of probe drugs for cytochrome P450 (CYP) isoenzymes (CYP1A2, CYP2C9, CYP2C19, CYP2D6, and CYP3A).

DETAILED DESCRIPTION:
Following a screening period, participants will receive DAC HYP over a 24-week treatment period (6 monthly injections) and then enter a 20-week washout period for assessment of immunogenicity, PK, pharmacodynamics, safety, and tolerability. The 20-week washout is necessary to ensure measurement of anti-DAC HYP binding antibodies (ADAbs) and neutralizing antibodies (NAbs) in the absence of drug interference. After washout, the participants may resume monthly treatment with DAC HYP 150 mg for an additional 3 years. All participants will be followed for 6 months after their last dose for safety monitoring. Additionally, two sub-studies will be performed: (1) an intensive serial PK sampling performed over the first and last dosing interval following DAC HYP doses administered at week 0 and at week 20, and (2) a therapeutic protein-drug interaction (TP-DI) sub-study, during which a probe drug cocktail will be administered at weeks 43 and 53 followed by serial probe-drug PK sampling up to 96 hours after probe-drug administration. A maximum of 20 participants will be enrolled in the TP-DI sub-study.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a confirmed diagnosis of RRMS according to McDonald criteria and previous cranial magnetic resonance imaging demonstrating lesion(s) consistent with MS
* Must have a baseline Expanded Disability Status Scale (EDSS) between 0.0 and 5.0, inclusive
* Must have had 1 or more clinical relapses within the previous 2 years
* Women of child bearing potential must be willing to practice effective contraception during the study and 4 months after the last dose

Key Exclusion Criteria:

* Other chronic disease of the immune system, malignancies, acute urologic, pulmonary, gastrointestinal disease
* Female subjects who are currently pregnant or breastfeeding

Key Inclusion criteria for 3-Year Treatment Extension:

To be eligible for participation in the 3-year treatment extension, participants must meet the following eligibility criteria at the time of reinitiation of DAC HYP:

* Must have been compliant with the 205MS302 (NCT01462318) protocol during the initial 24-week treatment period and the 20-week washout period in the opinion of the Investigator
* Must resume DAC HYP treatment ≤12 weeks after completion of the washout period (i.e., ≤12 weeks after their Week 44 visit).
* Participants who are currently receiving an approved IFN ß preparation must discontinue interferon (IFN) ß treatment at the time of reinitiation of DAC HYP dosing (no washout is required).

Key Inclusion criteria for the TP-DI Sub-study:

To be eligible for participation in the TP-DI Sub-Study, subjects must meet the following eligibility criteria at the Screening Visit at Week 40:

* Must have been compliant with the 205MS302 (NCT01462318) protocol during the initial 24-week treatment period and through Week 40 of the 20-week washout period in the opinion of the Investigator.
* Must agree to resume DAC HYP treatment ≤12 weeks after completion of the washout period (i.e., ≤12 weeks after their Week 44 visit).
* Must have normal liver function test results (total bilirubin ≤1.5 × upper limit of normal (ULN), alanine aminotransferase/aspartate aminotransferase ≤2 × ULN, and prothrombin time/partial thromboplastin time ≤1.2 × ULN).
* Must have normal renal function as estimated creatinine clearance >60 mL/min (Cockcroft-Gault formula).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (19):
- United States (7):
  - Research Site, Centennial, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Lake Barrington, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Farmington Hills, Michigan
  - Research Site, Dayton, Ohio
  - Research Site, Franklin, Tennessee
- Czechia (5):
  - Research Site, Brno
  - Research Site, Jihlava
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Teplice
- Hungary (5):
  - Research Site, Veszprém, Korhazu 1
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Székesfehérvár
- Poland (2):
  - Research Site, Katowice
  - Research Site, Krakow

REFERENCES:
- [Derived] Gold R, Stefoski D, Selmaj K, Havrdova E, Hurst C, Holman J, Tornesi B, Akella S, McCroskery P. Pregnancy Experience: Nonclinical Studies and Pregnancy Outcomes in the Daclizumab Clinical Study Program. Neurol Ther. 2016 Dec;5(2):169-182. doi: 10.1007/s40120-016-0048-2. Epub 2016 Jul 13. PMID 27411694

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Study: All participants received DAC HYP 150 mg SC injections every 4 weeks over an initial 24-week treatment period (for a total of 6 injections), followed by a 20-week washout period.
  Those participants from the Main Study who enrolled in the Intensive PK sub-study underwent serial DAC HYP PK sampling over the first and the last dosing intervals (on Day 1 [Week 0] and again on Day 141 [Week 20], the last dosing visit).
- Therapeutic Protein-Drug Interaction (TP-DI)Sub-study: In Period 1 (Week -1), the probe-drug cocktail (consisting of oral midazolam 5 mg, caffeine 200 mg, S-warfarin 10 mg, vitamin K 10 mg, omeprazole 40 mg, and dextromethorphan 30 mg, where the oral vitamin K was used prophylactically to counteract warfarin's anticoagulant effect) was administered 7 days before the first dose of DAC HYP 150 mg in the 3-year extension phase.
  In Period 2, pretreatment with DAC HYP 150 mg was administered at Weeks 0, 4, and 8. The probe-drug cocktail was administered 7 days after the third dose of DAC HYP.
- Extension Phase: After completion of the washout period from the Main Study or the TP-DI sub-study, eligible participants had the option to resume monthly open-label treatment with DAC HYP 150 mg in the extension phase of the study for up to 3 additional years.
Period: Main Study / TP-DI Study
Arm/Group | Main Study | Therapeutic Protein-Drug Interaction (TP-DI)Sub-study | Extension Phase
Started | 113 | 20 | 0
Enrolled in Intensive PK Substudy | 26 | 0 | 0
Completed | 105 | 20 | 0
Not Completed | 8 | 0 | 0
Not completed — Other | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0
Period: Extension Phase
Arm/Group | Main Study | Therapeutic Protein-Drug Interaction (TP-DI)Sub-study | Extension Phase
Started | 0 (95 participants from the Main Study entered the Extension Phase) | 0 (20 participants from the TP-DI Study entered the Extension Phase) | 115 (10 participants from the Main Study did not enter the Extension Phase.)
Completed | 0 | 0 | 70
Not Completed | 0 | 0 | 45
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1
Not completed — Disease Progression | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 15
Not completed — Investigator Decision | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 22

BASELINE CHARACTERISTICS:
Groups:
- TP-DI Sub-study: In Period 1 (Week -1), the probe-drug cocktail (consisting of oral midazolam 5 mg, caffeine 200 mg, S-warfarin 10 mg, vitamin K 10 mg, omeprazole 40 mg, and dextromethorphan 30 mg, where the oral vitamin K was used prophylactically to counteract warfarin's anticoagulant effect) was administered 7 days before the first dose of DAC HYP 150 mg in the 3-year extension phase.
  In Period 2, pretreatment with DAC HYP 150 mg was administered at Weeks 0, 4, and 8. The probe-drug cocktail was administered 7 days after the third dose of DAC HYP.
- Total: Total of all reporting groups
Arm/Group | Main Study | TP-DI Sub-study | Total
Number analyzed (Participants) | 113 | 20 | 133
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 0 | 0
  18 - 19 years | 0 | 1 | 1
  20 - 29 years | 28 | 4 | 32
  30 - 39 years | 40 | 7 | 47
  40 - 49 years | 31 | 5 | 36
  50 - 55 years | 14 | 3 | 17
  > 55 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 13 | 85
  Male | 41 | 7 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-DAC HYP Binding Antibodies (ADAbs): Electrochemiluminescent (ECL) Anti-Drug Antibody (ADA) Assay
Description: Participants with post-baseline (PB) ADAbs through Week 44, in the treatment period (extends up to 42 days after the last dose during the main study), and in the post-treatment period (43 days after the last dose until the end of the post-treatment period dose).
Time Frame: Up to 44 weeks
Population: Immunogenicity evaluable population: all participants in the main study population who received at least 1 dose of DAC HYP and had at least 1 post-study baseline immunogenicity assessment; n=participants with an assessment during the given period.
Measure: Number; unit: participants
Arm/Group | Main Study
Number analyzed (Participants) | 113
participants
  PB ADAbs through Week 44=negative; n=113 | 78
  PB ADAbs through Week 44=positive; n=113 | 35
  PB ADAbs in treatment period=negative; n=113 | 92
  PB ADAbs in treatment period=positive; n=113 | 21
  PB ADAbs in post-treatment period=negative; n=110 | 89
  PB ADAbs in post-treatment period=positive; n=110 | 21

2. Primary Outcome: Number of Participants With Anti-DAC HYP Neutralizing Antibodies (NAbs): ECL ADA Assay
Description: Participants with PB NAbs through Week 44, in the treatment period (extends up to 42 days after the last dose during the main study), and in the post-treatment period (43 days after the last dose until the end of the post-treatment period dose).
Time Frame: Up to 44 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Main Study
Number analyzed (Participants) | 113
participants
  PB NAbs through Week 44=negative; n=113 | 105
  PB NAbs through Week 44=positive; n=113 | 8
  PB NAbs in treatment period=negative; n=113 | 109
  PB NAbs in treatment period=positive; n=113 | 4
  PB NAbs in post-treatment period=negative; n=110 | 104
  PB NAbs in post-treatment period=positive; n=110 | 6

3. Primary Outcome: TP-DI Sub-study: Area-Under-the-Curve From Zero to Infinity (AUCinf) of Each Probe Drug
Description: AUCinf of each of the following cytochrome P450 (CYP) isoenzyme substrates: midazolam (CYP3A), S-warfarin + vitamin K (CYP2C9), and omeprazole (CYP2C19). The AUC from zero to 12 hours (AUC0-12) was calculated for caffeine (CYP1A2).
Time Frame: Week 43 (7 days prior to DAC HYP administration) and Week 53 (7 days after DAC HYP administration), pre-cocktail dose and at 0.5 and 1, 2, 3, 4, 6, 8, 10 , 24, 48, 72 and 96 hours post-probe drug cocktail administration
Population: TP-DI Sub-study population: all participants in the TP-DI substudy who had enough post-baseline measurable drug concentrations to calculate the parameter; n=participants with an evaluable assessment at given time point.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | TP-DI Sub-study
Number analyzed (Participants) | 20
hr*ng/mL
  Midazolam (Period 1) AUCinf; n=20 | 786.75 (328.794)
  Midazolam+DAC HYP (Period 2) AUCinf; n=19 | 816.87 (403.958)
  S-warfarin (Period 1) AUCinf; n=17 | 19292.9 (5524.60)
  S-warfarin+DAC HYP (Period 2) AUCinf; n=18 | 19609.3 (4620.64)
  Omeprazole (Period 1) AUCinf; n=18 | 2214.5 (2622.15)
  Omeprazole+DAC HYP (Period 2) AUCinf; n=19 | 1770.0 (1673.80)
  Caffeine (Period 1) AUC0-12; n=20 | 35742.4 (13942.71)
  Caffeine+DAC HYP (Period 2) AUC0-12; n=20 | 37449.2 (14367.04)
Statistical Analysis 1: Comparison: TP-DI Sub-study; Pairwise comparison: midazolam. Based on linear mixed model with fixed effect for treatment and random effect for participants; Test type: Superiority or Other; ratio = 1.015, 90% CI 2-sided [0.894 to 1.153] — test/reference = midazolam+DAC HYP/midazolam
Statistical Analysis 2: Comparison: TP-DI Sub-study; Pairwise comparison: S-warfarin. Based on linear mixed model with fixed effect for treatment and random effect for participants; Test type: Superiority or Other; ratio = 1.005, 90% CI 2-sided [0.951 to 1.063] — test/reference = S-warfarin+DAC HYP/S-warfarin
Statistical Analysis 3: Comparison: TP-DI Sub-study; Pairwise comparison: omeprazole. Based on linear mixed model with fixed effect for treatment and random effect for participants; Test type: Superiority or Other; ratio = 0.996, 90% CI 2-sided [0.880 to 1.127] — test/reference = omeprazole+DAC HYP/omeprazole
Statistical Analysis 4: Comparison: TP-DI Sub-study; Pairwise comparison: caffeine. Based on linear mixed model with fixed effect for treatment and random effect for participants. Excludes participants with high predose concentration (>5% of maximum observed concentration [Cmax]); Test type: Superiority or Other; ratio = 1.032, 90% CI 2-sided [0.930 to 1.145] — test/reference = caffeine+DAC HYP/caffeine

4. Primary Outcome: TP-DI Sub-study: Dextromethorphan to Dextrorphan Urine Concentration Ratio
Time Frame: Week 43 (7 days prior to DAC HYP administration) and Week 53 (7 days after DAC HYP administration), pre-cocktail dose and for 12 hours after probe-drug cocktail administration
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TP-DI Sub-study
Number analyzed (Participants) | 20
ratio
  Dextromethorphan (Period 1) | 0.42468 (1.258565)
  Dextromethorphan+DAC HYP (Period 2) | 0.48939 (1.813077)
Statistical Analysis 1: Comparison: TP-DI Sub-study; Pairwise comparison: dextromethorphan. Based on linear mixed model with fixed effect for treatment and random effect for participants; Test type: Superiority or Other; ratio = 1.012, 90% CI 2-sided [0.764 to 1.342] — test/reference = dextromethorphan+DAC HYP/dextromethorphan

5. Secondary Outcome: Intensive PK Sub-study: Cmax of DAC HYP
Time Frame: Day 1 and Day 141 (Week 20) at pre-dose and 8, 24, 72, and 120 hours post-dose and 7, 10, 14 and 21 days post-dose
Population: PK population: all participants who participated in the Intensive PK sub-study and had enough post-study baseline measurable drug concentrations to calculate the parameter; n=participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Main Study
Number analyzed (Participants) | 25
mcg/mL
  Day 1 (Week 0); n=25 | 12.63 (4.639)
  Day 141 (Week 20); n=24 | 29.07 (10.812)

6. Secondary Outcome: Intensive PK Sub-study: Time to Reach Maximum Concentration (Tmax) of DAC HYP
Time Frame: Day 1 and Day 141 (Week 20) at pre-dose and 8, 24, 72, and 120 hours post-dose and 7, 10, 14 and 21 days post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Main Study
Number analyzed (Participants) | 25
day
  Day 1 (Week 0); n=25 | 9.31 (6.368)
  Day 141 (Week 20); n=24 | 6.41 (3.273)

7. Secondary Outcome: Intensive PK Sub-study: Area-Under-the-Curve From Start to End of the Dosing Interval (AUCtau) of DAC HYP
Time Frame: Day 1 and Day 141 (Week 20) at pre-dose and 8, 24, 72, and 120 hours post-dose and 7, 10, 14, and 21 days post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Main Study
Number analyzed (Participants) | 25
day*mcg/mL
  Week 0 (Day 1); n=25 | 255.25 (88.569)
  Week 20; n=24 | 638.10 (256.076)

8. Secondary Outcome: Intensive PK Sub-study: Minimum Concentrations (Cmin) of DAC HYP
Time Frame: Day 141 (Week 20) at pre-dose and 8, 24, 72 and 120 hours post-dose and 7, 10, 14 and 21 days post-dose
Population: PK population: all participants who participated in the Intensive PK sub-study and had enough post-study baseline measurable drug concentrations to calculate the parameter.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Main Study
Number analyzed (Participants) | 24
mcg/mL | 14.93 (6.327)

9. Secondary Outcome: Intensive PK Sub-study: Apparent Volume of Distribution (V/F) of DAC HYP
Time Frame: Day 141 (Week 20) at pre-dose and 8, 24, 72 and 120 hours post-dose and 7, 10, 14 and 21 days post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Main Study
Number analyzed (Participants) | 24
Liters | 8.21 (2.810)

10. Secondary Outcome: Intensive PK Sub-study: Elimination Half-life (t½) of DAC HYP
Time Frame: Day 141 (Week 20) at pre-dose and 8, 24, 72 and 120 hours post-dose and 7, 10, 14 and 21 days post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Main Study
Number analyzed (Participants) | 24
day | 21.92 (5.473)

11. Secondary Outcome: Intensive PK Sub-study: Apparent Clearance (CL/F) of DAC HYP
Time Frame: Day 141 (Week 20) at pre-dose and 8, 24, 72 and 120 hours post-dose and 7, 10, 14 and 21 days post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | Main Study
Number analyzed (Participants) | 24
L/day | 0.27 (0.108)

12. Secondary Outcome: TP-DI Sub-study: Cmax of Each Probe Drug
Description: Cmax of each of the following CYP isoenzyme substrates: midazolam (CYP3A), caffeine (CYP1A2), warfarin + vitamin K (CYP2C9), and omeprazole (CYP2C19).
Time Frame: as for outcome 3
Population: TP-DI Substudy population: all participants in the TP-DI substudy who had enough post-baseline measurable drug concentrations to calculate the parameter; n=participants with an evaluable assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TP-DI Sub-study
Number analyzed (Participants) | 20
ng/mL
  Midazolam (Period 1); n=20 | 271.05 (106.925)
  Midazolam+DAC HYP (Period 2); n=19 | 311.21 (147.912)
  Caffeine (Period 1); n=20 | 4965.0 (1312.69)
  Caffeine+DAC HYP (Period 2); n=19 | 5399.5 (1364.05)
  S-Warfarin (Period 1); n=20 | 635.65 (140.291)
  S-Warfarin+DAC HYP (Period 2); n=19 | 649.74 (155.977)
  Omeprazole (Period 1); n=19 | 776.95 (513.344)
  Omeprazole+DAC HYP (Period 2); n=19 | 771.16 (540.331)
Statistical Analysis 1: Comparison: TP-DI Sub-study; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ratio = 1.079, 90% CI 2-sided [0.912 to 1.276] — test/reference = midazolam+DAC HYP/midazolam
Statistical Analysis 2: Comparison: TP-DI Sub-study; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; ratio = 1.012, 90% CI 2-sided [0.952 to 1.075] — test/reference = S-warfarin+DAC HYP/S-warfarin
Statistical Analysis 3: Comparison: TP-DI Sub-study; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; ratio = 1.058, 90% CI 2-sided [0.804 to 1.392] — test/reference = omeprazole+DAC HYP/omeprazole
Statistical Analysis 4: Comparison: TP-DI Sub-study; Pairwise comparison: caffeine. Based on linear mixed model with fixed effect for treatment and random effect for participants. Excludes participants with high predose concentration (>5% of Cmax); Test type: Superiority or Other; ratio = 1.116, 90% CI 2-sided [1.005 to 1.238] — test/reference = caffeine+DAC HYP/caffeine

13. Secondary Outcome: TP-DI Sub-study: CL/F of Each Probe Drug
Description: CL/F of each of the following CYP isoenzyme substrates: midazolam (CYP3A), warfarin + vitamin K (CYP2C9), and omeprazole (CYP2C19).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | TP-DI Sub-study
Number analyzed (Participants) | 20
mL/hr
  Midazolam (Period 1); n=20 | 7625.7 (3849.92)
  Midazolam+DAC HYP (Period 2); n=19 | 7298.6 (2844.22)
  S-Warfarin (Period 1); n=17 | 565.86 (184.129)
  S-Warfarin+DAC HYP (Period 2); n=18 | 541.46 (150.298)
  Omeprazole (Period 1); n=18 | 41612.4 (30003.48)
  Omeprazole+DAC HYP (Period 2); n=19 | 41772.4 (29810.30)

14. Secondary Outcome: TP-DI Sub-study: Omeprazole/Hydroxyomeprazole Concentration Ratio at 2 Hours Post-omeprazole Dosing
Time Frame: Week 43 (7 days prior to DAC HYP administration) and Week 53 (7 days after DAC HYP administration) at 2 hours after probe drug cocktail administration
Population: TP-DI Sub-study population: all participants in the TP-DI substudy who had enough post-baseline measurable drug concentrations to calculate the parameter.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TP-DI Sub-study
Number analyzed (Participants) | 17
ratio
  Omeprazole (Period 1) | 2.673 (4.7878)
  Omeprazole+ DAC HYP (Period 2) | 1.028 (0.9297)
Statistical Analysis 1: Comparison: TP-DI Sub-study; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; ratio = 0.878, 90% CI 2-sided [0.697 to 1.105] — test/reference = omeprazole+DAC HYP/omeprazole

ADVERSE EVENTS:
Time Frame: From Screening (for serious adverse events) or first dose of study treatment on Day 1 (for adverse events) through the end of treatment
Groups:
- DAC HYP 150 mg: DAC HYP 150 mg by SC injection using the PFS every 4 weeks for24 weeks followed by a 20-week washout period. After completion of the washout period, participants could resume monthly DAC HYP 150 mg using the PFS for up to 3 additional years. Participants in the TP-DI sub-study received s probe-drug cocktail administration at Weeks 43 and 53. The probe-drug cocktail consisted of midazolam 5 mg, caffeine 200 mg, S-warfarin 10 mg, vitamin K 10 mg, omeprazole 40 mg, and dextromethorphan 30 mg. The oral vitamin K was used to counteract warfarin's anticoagulant effect prophylactically.
Arm/Group | DAC HYP 150 mg
Serious Adverse Events (participants affected / at risk) | 33/133
Other Adverse Events (participants affected / at risk) | 106/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DAC HYP 150 mg (N=133)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Furuncle (Infections and infestations) | 1
Hepatitis E (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Streptococcal urinary tract infection (Infections and infestations) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Obesity (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 10
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2
Cutaneous sarcoidosis (Skin and subcutaneous tissue disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DAC HYP 150 mg (N=133)
Lymphadenopathy (Blood and lymphatic system disorders) | 8
Hypothyroidism (Endocrine disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 12
Influenza like illness (General disorders) | 13
Pyrexia (General disorders) | 12
Influenza (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 19
Oral herpes (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 15
Sinusitis (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 33
Urinary tract infection (Infections and infestations) | 30
Alanine aminotransferase increased (Investigations) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Spinal pain (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 21
Hypoaesthesia (Nervous system disorders) | 9
Migraine (Nervous system disorders) | 7
Multiple sclerosis relapse (Nervous system disorders) | 58
Muscle spasticity (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.